CLINICAL TRIAL: NCT01111838
Title: A Phase II Clinical and Translational Study of STA-9090 in Patients With Refractory Metastatic Colorectal Cancer
Brief Title: Clinical and Translational Study of STA-9090
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-029
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: STA-9090; colon; rectal; 10-029
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — STA 9090

ARMS (1):
- STA-9090 (Experimental): This is an open-label Phase 2 clinical study in patients with advanced colorectal cancer (CRC). Patients will be treated with 200mg/m2 of STA-9090 during a 1-hour intravenous infusion 1 time per week for three consecutive weeks followed by a 1 week dose-free interval. Patients tolerating STA-9090 will be permitted to continue treatment until disease progression.
  Interventions: Drug: STA-9090

INTERVENTIONS:
Drug: STA-9090 — Patients will be enrolled and receive 200mg/m2 of STA-9090. Patients will receive single agent STA-9090 intravenous (I.V.) infusion (an indwelling catheter may not be used) over 60 minutes weekly (three weeks on and one week off). Follow-up imaging will be performed every 8 weeks to evaluate response.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad STA-9090 has on colorectal cancer. This is a phase II trial which tests both how well the drug works in fighting your cancer as well as any possible side effects it will have on the patient.

Cancer is a disease of uncontrolled growth. This growth is controlled in part by a series of proteins that are part of a growth pathway. Some of these proteins are destroyed by a protein called HSP90 and STA-9090 is a test drug which blocks one of the proteins that helps cancer grow. This study will also look at molecular markers that may affect how the cancer grows, and how it responds to treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has histologically or cytologically-confirmed colorectal cancer with metastatic disease documented on diagnostic imaging studies.
* The patient has measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded), measuring ≥20 mm on conventional measurement techniques or ≥10 mm on spiral computed tomography (CT) scan.
* The patient has received at least one prior standard and/or investigational regimen for metastatic disease.
* The patient is age ≥18 years.
* The patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1 (Karnofsky≥ 80%).
* The patient has adequate hematologic function as defined by an absolute neutrophil count ≥1500/μL, hemoglobin ≥9/μdL, and a platelet count ≥100,000/μL.
* The patient has adequate hepatic function as defined by a total bilirubin ≤ 2.5x the upper limit of normal (ULN), and aspartate transaminase (AST) and alanine transaminase (ALT)≤3 x the ULN (or ≤5 x the ULN in the presence of known liver metastases).
* The patient, if not on anticoagulation, has adequate coagulation function as defined by international normalized ratio (INR) ≤1.5 ULN and partial thromboplastin time (PTT) ≤1.5x the ULN. Patients on full-dose anticoagulation must be on a stable dose of oral anticoagulation or low molecular weight heparin, must have an INR value within acceptable range for treatment and have no active bleeding or pathological condition that, in the opinion of the investigator, carries a high risk of bleeding.
* The patient has adequate renal function as defined by serum creatinine ≤1.5 x the institutional ULN or creatinine clearance ≥60 mL/min for patients with creatinine levels above 1.5, as well as urine protein ≤1+ on routine analysis (if routine UA indicates ≥2+ protein, a 24-hour urine collection for protein must demonstrate < 1000mg of protein in 24 hours to allow participation in the study).
* The patient has a life expectancy of > 3 months.
* Because the teratogenicity of STA-9090 is not known, men and women of childbearing potential must agree to use adequate contraception (hormonal or barrier birth control; abstinence) prior to study entry and for the duration of study participation.
* The patient has the ability to read and willingness to sign informed consent.
* For stage I of the protocol (the first 15 patients) the tumor must be amenable to biopsy and the patient must be willing to undergo pre and post treatment biopsies.
* The patient must have a normal QTc interval on baseline ECG , (<470 milliseconds, males and females).

Exclusion Criteria:

* Patient may not have received chemotherapy within 4 weeks prior to entering the study, and must have recovered (to grade 1 or less) from adverse events due to agents administered.
* Primary brain tumors or active brain metastases. However, patients with a history of CNS metastases will be eligible if they have been treated and are stable for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on a stable dose of steroids for a minimum of 2 weeks prior to enrollment.
* History of stroke within 6 months of treatment or other significant neurological limitations.
* Major surgery within 4 weeks prior to entering the study.
* Poor venous access for study drug administration or would require a peripheral or central indwelling catheter for study drug administration. Study drug administration via indwelling catheters is prohibited at this time.
* Use of any investigational agents within 4 weeks prior to entering the study.
* History of severe allergic reactions to excipients (e.g., Polyethylene glycol 300 and Polysorbate 80), including severe hypersensitivity reactions defined as ≥ Grade 3 based on NCI CTCAE version 3.
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation or systemic steroids for treatment of autoimmune disease). However, patients may receive steroids for stable CNS metastases as described in exclusion criterion 2.
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive patients receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Ventricular ejection fraction (Ef) ≤ 45%.
* Inaccessible tissue for biopsy (first 15 patients only)
* History of or current coronary artery disease, myocardial infarction, angina pectoris, angioplasty or coronary bypass surgery
* History of or current uncontrolled dysrhythmias, or requirement for antiarrhythmic medications, or Grade 2 or greater left bundle branch block
* New York Heart Association class II/III/IV congestive heart failure with a history of dyspnea, orthopnea or edema that requires current treatment with angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, beta-blockers or diuretics
* Current or prior radiation therapy to the left hemithorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Refractory Metastatic Colorectal Cancer: Clinical and Translational Study of STA-9090 in Patients with Refractory Metastatic Colorectal Cancer
Period: Overall Study
Arm/Group | Patients With Refractory Metastatic Colorectal Cancer
Started | 22
Completed | 15
Not Completed | 7
Not completed — Patient Ineligible | 2
Not completed — Not Treated | 3
Not completed — Clinical deterioration | 1
Not completed — Other Complicating Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Refractory Metastatic Colorectal Cancer
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: To Determine Overall Objective Response.
Description: Patients with measurable disease will be evaluated using RECIST criteria for determination of response.
Time Frame: every 8 weeks
Measure: Number; unit: participants
Arm/Group | Patients With Refractory Metastatic Colorectal Cancer
Number analyzed (Participants) | 15
participants
  Progression of Disease (POD) | 9
  Stable Disease (SD) | 6

ADVERSE EVENTS:
Arm/Group | Patients With Refractory Metastatic Colorectal Cancer
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Refractory Metastatic Colorectal Cancer (N=15)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Amylase (Blood and lymphatic system disorders) | 1 (1)
Ascites (non-malignant) (General disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Renal and urinary disorders) | 2 (2)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1)
Lipase (Metabolism and nutrition disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Neurology - Other (specify) (Nervous system disorders) | 1 (1)
Obstruction, GI- Colon (Gastrointestinal disorders) | 1 (1)
Obstruction, GI- Small bowel NOS (Gastrointestinal disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 2 (2)
Vomiting (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Refractory Metastatic Colorectal Cancer (N=15)
ALT, SGPT (Blood and lymphatic system disorders) | 7 (7)
AST, SGOT (Blood and lymphatic system disorders) | 9 (9)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6 (6)
Alkaline phosphatase (Metabolism and nutrition disorders) | 10 (10)
Allergy reaction (including drug fever) (General disorders) | 1 (2)
Amylase (Blood and lymphatic system disorders) | 4 (4)
Anorexia (Psychiatric disorders) | 3 (4)
Ascites (non-malignant) (General disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 6 (6)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1)
Constitutional Symptoms (General disorders) | 2 (2)
Dental: dentures or prosthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (14)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (12)
Fever (in the absence of neutropenia) (General disorders) | 2 (2)
Gastrointestinal, other (Gastrointestinal disorders) | 1 (1)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 7 (7)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5)
INR (Blood and lymphatic system disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (3)
Lipase (Metabolism and nutrition disorders) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 6 (6)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Metabolic/Lab (Metabolism and nutrition disorders) | 2 (2)
Nausea (General disorders) | 4 (4)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (3)
Obstruction, GI- Small bowel NOS (Gastrointestinal disorders) | 1 (1)
PTT (Blood and lymphatic system disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 4 (4)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 5 (5)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 3 (3)
Sweating (diaphoresis) (General disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vomiting (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes